CLINICAL TRIAL: NCT01969084
Title: The Effect of Linagliptin on Mitochondrial and Endothelial Function
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Aristidis Veves, Research Director, Microcirculation Lab and Joslin-Beth Israel Deaconess Foot Center, Beth Israel Deaconess Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2013P-000057; IIS trial 1218.137 (Other Grant/Funding Number: BIPI)
Record Dates: First submitted 2013-08-29; First posted 2013-10-25 (Estimated); Results first posted 2016-11-18 (Estimated); Last update posted 2016-11-18 (Estimated); Status verified 2016-11

CONDITIONS: Type II Diabetes Mellitus
Keywords: Type II Diabetes Mellitus; Diabetes; Metabolism; Linagliptin; Tradjenta; Glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus | interventions — Linagliptin; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Linagliptin (Experimental): Subjects given Linagliptin
  Interventions: Drug: Linagliptin; Other: Microcirculation testing; Other: Macrocirculation testing; Other: MRI Scans
- Sugar pill (Placebo Comparator): Subjects given sugar pill/placebo
  Interventions: Drug: Placebo; Other: Microcirculation testing; Other: Macrocirculation testing; Other: MRI Scans

INTERVENTIONS:
Drug: Linagliptin
  Other Names: Tradjenta
  Arms: Linagliptin
Drug: Placebo
  Arms: Sugar pill
Other: Microcirculation testing — The endothelial function of the micro-circulation will be assessed by measuring the hyperemic response of the vessels in the superficial skin of the forearm after the iontophoresis of acetylcholine. The endothelium independent vasodilation will be assessed by the iontophoresis of sodium nitroprusside. Laser Doppler perfusion imaging will be used to measure relative changes in flow velocity.Visible and NIR Medical Hyperspectral Imaging (MHSI) data will be collected with a HyperMed OxyView MHSI System (HyperMed, Inc., Watertown, MA). MHSI images will be obtained from same forearm area where the iontophoresis of acetylcholine and sodium nitroprusside will be performed, before and after the iontophoresis test.
Other: Macrocirculation testing — Use ultrasound to measure brachial artery flow mediated vasodilation (FMD, endothelium-dependent vasodilation) and nitroglycerin induced dilation (NID, endothelium-independent vasodilation).
Other: MRI Scans — Phosphorus-31 MRI data will be obtained during an exercise protocol. Muscle oxygenation will be measured using the blood oxygenation level-dependent magnetic resonance imaging (BOLD MRI) technique after induced hyperemia.

SUMMARY:
Investigators propose to examine the effect of 12 weeks of Linagliptin, a diabetes drug, treatment on inflammation as well as vascular and mitochondrial function in diabetic patients. Investigators hypothesize that Linagliptin will reduce the proinflammatory state, improve endothelial function, increase the blood flow at the muscle microcirculation level and improve mitochondrial function. In this study, investigators will perform tests that evaluate the function of small and large blood vessels by employing ultrasound and laser doppler techniques. In addition MRI scans that evaluate the mitochondrial function of the lower extremity muscles at rest and during exercise will also be employed. Forty subjects with Type 2 diabetes will be studied for twelve weeks and half of them will be randomly assigned to receive linagliptin while the other half will receive placebo. All tests will be performed at the beginning and the end of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients with T2DM whose medical or lifestyle treatment regimen is stable and not expected to be changed during the study period. Patients will be considered stable on their treatment regimen if there have not been any changes in the type of their antidiabetic medications over the past 3 months and/or there have not been any changes in their blood glucose levels that have caused them to see their health care provider more often than usual over the preceding three months. The diagnosis of T2DM will be according to the American Diabetes Association criteria. Subjects previously diagnosed with T2DM will not require confirmatory testing.
* Age 30-70 years
* Patients on insulin should be on a stable insulin regimen for at least 4 months prior to enrollment.
* Patients on antidiabetic treatment will be eligible if they are stable and no change in their treatment is planned for the next three months while they are in the study.
* HBA1c ≤ 10.0

Exclusion Criteria:

* Patient with unstable diabetes that has resulted in hyperosmolar coma, DKA, and/or documented increase or decrease in HbA1c of more than 2.0% within the previous 6 months
* Treatment with DPP4 Inhibitors or GLP-1 agonists. Patients who discontinued such treatment should be at least free for a 3-month period.
* Severe proliferative retinopathy that renders the subject legally blinded
* Previously intermittent claudication or diagnosed severe peripheral arterial disease requiring intervention.
* History of Deep Vein Thrombosis (DVT) within the past 3 months.
* Significant limb swelling due to lymphedema
* Previous diagnosis of severe gastroparesis diabeticorum due to autonomic neuropathy that has necessitated hospital admission
* Presence of non-healing foot ulceration due to severe peripheral diabetic neuropathy
* History of pancreatitis
* Documented diabetic nephropathy manifested as macro-albuminuria before enrollment in the study, (2 of 3 urine specimens collected within a 3-6 month period with urine albumin> 300 ug/mg creatinine - according to the ADA position statement)
* Smokers. Smokers will be defined as any subject who reports tobacco use during the three months before to study enrollment.
* Active or uncontrolled cardiovascular disease as follows:

  1. Myocardial infarction, or angina within 12 months of study participation
  2. Arrhythmia (uncontrolled, highly symptomatic, requires treatment or life-threatening).
  3. Patients with congestive heart failure requiring pharmacologic management, particularly when accompanied by hypoperfusion and hypoxemia due to unstable or acute failure, are at increased risk of lactic acidosis.
  4. Stroke or transient ischemic attack within 12 months of study participation
  5. Uncontrolled hypertension: SBP> 180 mmHg or DBP> 105 mmHg (2 abnormal readings during visit)
* Liver disease (AST, ALT Alk Phos levels >2x upper normal limit) at the time of enrollment
* Renal disease (creatinine > 2 mg/dL and/or estimated GFR <30 mL/min, history of dialysis, nephrotic syndrome) at the time of enrollment.
* Severe dyslipidemia (triglycerides>600 mg/dL or cholesterol >350 mg/dL) Subjects with hypertriglyceridemia may be retested in 2-3 weeks as the values can fluctuate tremendously within a few days. In the event that the retested value allows the patient to be enrolled, a planned deviation will be submitted to the CCI.
* Any other serious chronic disease requiring active treatment.
* Pregnancy or Lactation
* Females of childbearing potential not using an effective form of birth control as determined by the investigators.
* Subjects on any of the following medications:

  1. Systemic (not inhaled) Glucocorticoids
  2. Antineoplastic agents
  3. Rifampin
* Patient is known to have a history of immunodeficiency diseases, including a positive HIV (ELISA and Western blot) and/or positive Hepatitis B surface antigen (HBsAg) or Hepatitis C test result in the past.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or baseline evaluations.
* Acute or chronic metabolic acidosis, including diabetic ketoacidosis.
* History of hypersensitivity reaction to linagliptin (such as urticaria, angioedema, or bronchial hyperreactivity) or metformin.
* Contraindications to MRI: Medically unstable or hematologic, renal, or hepatic dysfunction, cardiac pacemaker, Intracranial clips, metal implants, or external clips within 10 mm of the head,
* Metal in eyes.
* Pregnant or nursing women -
* Claustrophobia.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2013-10; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

REFERENCES:
- [Result] Baltzis D, Dushay JR, Loader J, Wu J, Greenman RL, Roustit M, Veves A. Effect of Linagliptin on Vascular Function: A Randomized, Placebo-controlled Study. J Clin Endocrinol Metab. 2016 Nov;101(11):4205-4213. doi: 10.1210/jc.2016-2655. Epub 2016 Sep 1. PMID 27583476

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 45 subjects were enrolled and 41 were randomized to the study
Groups:
- Linagliptin: Subjects given Linagliptin
  Linagliptin
  Microcirculation testing: The endothelial function of the micro-circulation was assessed by measuring the hyperemic response of the vessels in the superficial skin of the forearm after the iontophoresis of acetylcholine. The endothelium independent vasodilation will be assessed by the iontophoresis of sodium nitroprusside. Laser Doppler perfusion imaging will be used to measure relative changes in flow velocity.Visible and NIR Medical Hyperspectral Imaging (MHSI) data will be collected with a HyperMed OxyView MHSI System (HyperMed, Inc., Watertown, MA). MHSI images will be obtained from same forearm area where the iontophoresis of acetylcholine and sodium nitroprusside will be performed, before and after the iontophoresis test.
  Macrocirculation testing: Use ultrasound to measure brachial artery flow mediated vasodilation (FMD, endothelium-dependent vasodilation) and nitroglycerin induced dilation (NID, endothelium-independent vasodila
- Sugar Pill: Subjects given sugar pill/placebo
  Placebo
  Microcirculation testing: The endothelial function of the micro-circulation was assessed by measuring the hyperemic response of the vessels in the superficial skin of the forearm after the iontophoresis of acetylcholine. The endothelium independent vasodilation will be assessed by the iontophoresis of sodium nitroprusside. Laser Doppler perfusion imaging will be used to measure relative changes in flow velocity.Visible and NIR Medical Hyperspectral Imaging (MHSI) data will be collected with a HyperMed OxyView MHSI System (HyperMed, Inc., Watertown, MA). MHSI images will be obtained from same forearm area where the iontophoresis of acetylcholine and sodium nitroprusside will be performed, before and after the iontophoresis test.
  Macrocirculation testing: Use ultrasound to measure brachial artery flow mediated vasodilation (FMD, endothelium-dependent vasodilation) and nitroglycerin induced dilation (NID, endothelium-independent vasod
Period: Overall Study
Arm/Group | Linagliptin | Sugar Pill
Started | 19 | 22
Completed | 19 | 21 (One subject withdrew due to unrelated serious adverse event)
Not Completed | 0 | 1
Not completed — Adverse Event | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Linagliptin | Sugar Pill | Total
Number analyzed (Participants) | 19 | 22 | 41
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 20 | 34
  >=65 years | 5 | 2 | 7
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.79 (5.75) | 56.76 (6.79) | 58.67 (6.56)
Gender [Count of Participants; unit: Participants]
  Female | 7 | 11 | 18
  Male | 12 | 11 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 19 | 22 | 41

OUTCOME MEASURES:

1. Primary Outcome: Phosphocreatine (PCR) Recovery Time After Exhaustive or up to 6 Minutes of Leg Exercise.
Description: Change in the time to phosphocreatine recovery between the baseline visit and post-treatment visit following the graded exercise test.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: seconds
Groups:
- Linagliptin: Subjects given Linagliptin
  Linagliptin
  MRI Scans: Phosphorus-31 MRI data was obtained during an exercise protocol. Muscle oxygenation will be measured using the blood oxygenation level-dependent magnetic resonance imaging (BOLD MRI) technique after induced hyperemia.
- Sugar Pill: Subjects given sugar pill/placebo
  Placebo
  MRI Scans: Phosphorus-31 MRI data was obtained during an exercise protocol. Muscle oxygenation will be measured using the blood oxygenation level-dependent magnetic resonance imaging (BOLD MRI) technique after induced hyperemia.
Arm/Group | Linagliptin | Sugar Pill
Number analyzed (Participants) | 19 | 21
seconds | 0.0 [-23.3 to 15.3] | 1.01 [-36.8 to 14.0]
Statistical Analysis 1: Comparison: Linagliptin vs Sugar Pill; Data were expressed as the median (25th:75th percentiles) for non-normally distributed data. The mean±sd for the groups was not analyzed as per the statistical plan; Test type: Superiority or Other; p > 0.05, Wilcoxon (Mann-Whitney) — A p-value of < 0.05 was considered statistically significant

2. Secondary Outcome: Change in Muscle Oxygenation Recovery Time
Description: Change in muscle oxygenation after ischemia inducing occlusion for 4 minutes.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: seconds
Arm/Group | Linagliptin | Sugar Pill
Number analyzed (Participants) | 19 | 21
seconds
  Medial gastrocnemius | 2.6 [-6.2 to 13.9] | 7.1 [-7.1 to 10.1]
  Lateral gastrocnemius | 2.8 [-6.6 to 11.3] | 2.2 [-9.1 to 8.1]
  Soleus | 0.3 [-3.6 to 3.9] | -1.6 [-3.9 to 2.2]
  Tibialis anterior | 2.9 [1.2 to 27.1] | 2.40 [-6.6 to 8.6]
  Peroneus Longus | 0.4 [-4.0 to 7.1] | -0.12 [-2.0 to 2.6]

3. Secondary Outcome: Changes in Vascular Reactivity in the Micro- and Macro-circulation.
Description: Change in markers of macro- and microvascular function from the baseline visit to the post-treatment visit between the two groups.
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: percent change
Groups:
- Linagliptin: Linagliptin treated group
- Sugar Pill: Subjects given sugar pill/placebo
  Placebo
  Microcirculation testing: The endothelial function of the micro-circulation was assessed by measuring the hyperemic response of the vessels in the superficial skin of the forearm after the iontophoresis of acetylcholine. The endothelium independent vasodilation will be assessed by the iontophoresis of sodium nitroprusside. Laser Doppler perfusion imaging will be used to measure relative changes in flow velocity
Arm/Group | Linagliptin | Sugar Pill
Number analyzed (Participants) | 19 | 21
percent change
  ACh LDPI | 14.2 [-9.5 to 25.4] | -6.1 [-15.3 to 22.6]
  ACh axon reflex | 48.5 [-47.8 to 125.7] | -7.4 [-259.2 to 153.2]
  Flow mediated dilation | 0.67 [-0.58 to 1.58] | 0.36 [-0.38 to 1.21]
  Nitroglycerin mediated dilation | 0.27 [-0.78 to 1.62] | 0.11 [-0.91 to 1.21]

4. Secondary Outcome: Changes in SDF1-α and Substance P
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Linagliptin | Sugar Pill
Number analyzed (Participants) | 19 | 21
pg/ml
  SDF-1 | 3 [-100 to 28] | 11.1 [-1.2 to 53]
  Substance P | 77.4 [-69.7 to 348.0] | 42.2 [-349.0 to 138.8]

5. Secondary Outcome: Changes in Circulating Endothelial Progenitor Cell Phenotypes
Description: The measurements of the various EPC phenotypes were performed at the Beth Israel Deaconess Flow Cytometry Core Facility. Immunofluorescent cell staining was performed on peripheral blood with the use of the fluorescent conjugated antibodies. 1.000.000 events per sample were acquired using a FACS LSR II analyzer (Becton Dickinson, Franklin Lakes, NJ, USA) and the results were analyzed using the Beckman Coulter Kaluza analysis software (Beckman Coulter Inc., Brea, CA, USA).
Time Frame: Baseline and 12 weeks
Measure: Median (Inter-Quartile Range); unit: Events per million
Arm/Group | Linagliptin | Sugar Pill
Number analyzed (Participants) | 19 | 21
Events per million
  CD133-KDR | 5 [-20 to 111] | 1 [-45 to 40]
  KDR-CD34 | 1 [-26 to 74] | 1 [-15 to 49]
  CD133-CD34-KDR | 4 [-4 to 102] | -3 [-15 to 5]

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: whole study period
Groups:
- Sugar Pill: Subjects given sugar pill/placebo
  Placebo
Arm/Group | Linagliptin | Sugar Pill
Serious Adverse Events (participants affected / at risk) | 1/19 | 3/22
Other Adverse Events (participants affected / at risk) | 2/19 | 4/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin (N=19) | Sugar Pill (N=22)
Leg blisters (Skin and subcutaneous tissue disorders) | 1 (1) | 0 — Blisters on legs
acute kidney injury (Renal and urinary disorders) | 0 | 1
Car accident (Social circumstances) | 0 | 1
Decreased eGFR (Renal and urinary disorders) | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Linagliptin (N=19) | Sugar Pill (N=22)
Increased creatinine and BUN, reduced GFR (Renal and urinary disorders) | 1 | 3
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cramping in the calf muscle during the graded exercise test (Musculoskeletal and connective tissue disorders) | 0 | 1 (1)
Decreased CO2 concentration (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Lung water accumulation (Respiratory, thoracic and mediastinal disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No